CLINICAL TRIAL: NCT01322568
Title: Age, Gene/Environment Susceptibility (AGES) Study
Brief Title: Research on Aging Project in Iceland: Second Stage
Status: Completed | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999903319; 03-AG-N319
Record Dates: First submitted 2011-03-23; First posted 2011-03-24 (Estimated); Last update posted 2019-11-12 (Actual); Status verified 2014-02-11

CONDITIONS: Atherosclerosis; Osteoporosis; Obesity; Glucose Abnormalities; Alzheimer's Disease; Vascular Dimentia
Keywords: Aging; Gene; Environment; Inflammation; Iceland
MeSH Terms: conditions — Atherosclerosis; Osteoporosis; Obesity; Alzheimer Disease; Inflammation

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Researchers are interested in studying the environmental and genetic factors that play a role in health and living conditions as people age. Since 2002, the U.S. National Institute on Aging and the Icelandic Heart Association Research Institute have been conducting a long-term study known as the Research in Aging project to collect personal data and samples from Icelandic men and women in order to study risk factors related to disease and disability in old age. Researchers plan to initiate a second stage of the study.

Objectives:

- To collect additional personal information, medical records, and blood samples from individuals who have previously provided materials for the Research in Aging Project in Iceland.

Eligibility:

- Individuals who have previously participated in the Research in Aging project in association with the U.S. National Institute on Aging and the Icelandic Heart Association Research Institute.

Design:

* Participants will have a physical examination with imaging analysis procedures and hearing and eye tests, provide information on health and diet, and provide a 100-ml blood sample for testing.
* Participants will also provide consent for researchers to consult data and samples collected during the first stage of the Research on Aging project.

DETAILED DESCRIPTION:
In anticipation of the sequencing of the human genome and description of the human proteome, the Age, Gene/Environment Susceptibility-Reykjavik Study (AGES) was initiated in 2002. AGES was designed to examine risk factors, including genetic susceptibility and gene/environment interaction, in relation to disease and disability in old age. The study is multidisciplinary, providing detailed phenotypes related to the cardiovascular, neurocognitive (including sensory), and musculoskeletal systems, and to body composition and metabolic regulation. Relevant quantitative traits, subclinical indicators of disease, and medical diagnoses are identified by using biomarkers, imaging, and other physiologic indicators. The AGES sample is drawn from an established population-based cohort, the Reykjavik Study. This cohort of men and women born between 1907 and 1935 has been followed in Iceland since 1967 by the Icelandic Heart Association. The AGES cohort, with cardiovascular risk factor assessments earlier in life and detailed late- life phenotypes of quantitative traits, will create a comprehensive study of aging nested in a relatively genetically homogeneous older population. This approach should facilitate identification of genetic factors that contribute to healthy aging as well as the chronic conditions common in old age.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals who have previously participated in the Research in Aging project in association with the U.S. National Institute on Aging and the Icelandic Heart Association Research Institute.

Ages: 32 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5764 (Actual)
Dates: Start 2003-01-31; Study Completion 2014-02-11

CONTACTS AND LOCATIONS:
Overall Officials: Tamara B Harris, M.D., Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- Icelandic Heart Association Research Institute, Kopavogur, Iceland

REFERENCES:
- [Background] Freimer N, Sabatti C. The human phenome project. Nat Genet. 2003 May;34(1):15-21. doi: 10.1038/ng0503-15. No abstract available. PMID 12721547
- [Background] Ross R. Atherosclerosis--an inflammatory disease. N Engl J Med. 1999 Jan 14;340(2):115-26. doi: 10.1056/NEJM199901143400207. No abstract available. PMID 9887164
- [Background] Ershler WB, Keller ET. Age-associated increased interleukin-6 gene expression, late-life diseases, and frailty. Annu Rev Med. 2000;51:245-70. doi: 10.1146/annurev.med.51.1.245. PMID 10774463
- [Derived] Schelbert EB, Cao JJ, Sigurdsson S, Aspelund T, Kellman P, Aletras AH, Dyke CK, Thorgeirsson G, Eiriksdottir G, Launer LJ, Gudnason V, Harris TB, Arai AE. Prevalence and prognosis of unrecognized myocardial infarction determined by cardiac magnetic resonance in older adults. JAMA. 2012 Sep 5;308(9):890-6. doi: 10.1001/2012.jama.11089. PMID 22948699